CLINICAL TRIAL: NCT03037853
Title: Anatomic Altas of the Whole Human Body
Acronym: A2H
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: A2H
Record Dates: First submitted 2016-07-08; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteer
Keywords: Atlas; Full human Body; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy volunteers: Healthy volunteers
  Interventions: Other: Healthy volunteers

INTERVENTIONS:
Other: Healthy volunteers — MRI scanner

SUMMARY:
The goal is the constitution of a statistical atlas of the human being morphology variability.

This work would be a significant step forward in the field of anatomy and biomechanical simulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18 and 99 years.

Exclusion Criteria:

* Respiratory and cardiovascular pathology
* Claustrophobia
* Counter-argument to magnetic field exposure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers adults.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Constitution of a statistical atlas of the full human body | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Palombi, Professor, Principal Investigator — Grenoble Hospital University

REFERENCES:
- [Background] Palombi O, Ulliana F, Favier V, Leon JC, Rousset MC. My Corporis Fabrica: an ontology-based tool for reasoning and querying on complex anatomical models. J Biomed Semantics. 2014 May 6;5:20. doi: 10.1186/2041-1480-5-20. eCollection 2014. PMID 24936286
- [Background] Anatomy Transfer Ali Hamadi Dicko; Tiantian Liu; Benjamin Gilles; Ladislav Kavan; François Faure; Olivier Palombi; Marie-Paule Cani ACM Transactions on Graphics, ACM, 2013, ACM SIGGRAPH ASIA, 32 (6), pp. Article No. 188
- [Background] Frame-based interactive simulation of complex deformable objects Benjamin Gilles; François Faure; Guillaume Bousquet; Dinesh K. Pai Deformation Models, 7, Springer, pp. 145-166, 2013, Lecture Notes in Computational Vision and Biomechanics, 978-94-007-5446-1
- [Background] SOFA: A Multi-Model Framework for Interactive Physical Simulation François Faure; Christian Duriez; Hervé Delingette; Jérémie Allard; Benjamin Gilles; Stéphanie Marchesseau; Hugo Talbot; Hadrien Courtecuisse; Guillaume Bousquet; Igor Peterlik; Stéphane Cotin. In Yohan Payan. Soft Tissue Biomechanical Modeling for Computer Assisted Surgery, 11, Springer, pp. 283-321, Jun. 2012, Studies in Mechanobiology, Tissue Engineering and Biomaterials, 978-3-642-29013-8
- [Background] From Generic to Specic Musculoskeletal Simulations using an Ontology-based Modeling Pipeline Ali Hamadi Dicko; Benjamin Gilles; François Faure; Olivier Palombi Dimitri Plemenos and Georges Miaoulis. Intelligent Computer Graphics 2012, 441, Springer, pp. 227-242, May. 2012, Studies in Computational Intelligence
- [Background] Doppler Ultrasound Driven Biomechanical Model of the Brain for Intraoperative Brain-Shift Compensation: A Proof of Concept in Clinical Conditions Marek Bucki; Olivier Palombi; Mathieu Bailet; Yohan Payan Yohan Payan. Soft Tissue Biomechanical Modeling for Computer Assisted Surgery, Springer-Verlag, pp. 135-165, 2012, Studies in Mechanobiology, Tissue Engineering and Biomaterials, 978-3-642-29013-8
- [Background] Statistical models of appearance for medical image analysis and computer vision, in medical imaging. T.F. Cootes and C.J. Taylor. Proc. of SPIE, 4322:238-248, 2001.
- [Background] Creating and animating subject-specific anatomical models, B. Gilles, L. Revéret, D.K. Pai Computer Graphics Forum, presented at Eurographics'11, 29(8), pp 2340-2351, 2010.